CLINICAL TRIAL: NCT00372996
Title: A Two-arm Randomized Open Label Phase 2 Study Of Cp-751,871 In Combination With Exemestane Versus Exemestane Alone As First Line Treatment For Postmenopausal Patients With Hormone Receptor Positive Advanced Breast Cancer
Brief Title: Study Of CP-751,871 In Combination With Exemestane In Postmenopausal Women With Hormone Receptor Positive Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed to enrollment as of 13 May 2011 due to business reasons. Premature closure was not prompted by any safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021004; 2006-005573-21 (EudraCT Number)
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — figitumumab; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CP-751,871 + exemestane Treatment until progression or toxicity
  Interventions: Drug: CP-751,871; Drug: exemestane; Drug: Fulvestrant
- 2 (Active Comparator)
  Interventions: Drug: exemestane

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 given at 20 mg/kg IV on day 1 of each 21 day cycle.
  Arms: 1
Drug: exemestane — Exemestane given at 25 mg orally once a day.
  Arms: 1
Drug: exemestane — Exemestane given at 25 mg orally once a day. Treatment until progression or toxicity
  Arms: 2
Drug: Fulvestrant — Used for salvage therapy and administered according to the local label and standard clinical practice.
  Arms: 1

SUMMARY:
To test the efficacy of CP-751,871 combined with exemestane in the treatment of postmenopausal patients with hormone positive advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with a diagnosis of hormone receptor positive advanced breast cancer
* HbA1c <5.7%

Exclusion Criteria:

* Previous treatment for advanced disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (31):
  - UCSD Medical Center - La Jolla, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - Washington Cancer Institute (WCI) at Washington Hospital Center (WHC), Washington D.C., District of Columbia
  - Florida Cancer Research Institute, Davie, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Central Baptist Hospital, Lexington, Kentucky
  - Lexington Oncology Associates, Lexington, Kentucky
  - Bluegrass Hematology/Oncology, PSC, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of Minnesota Medical Center-Fairview, Riverside Campus, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University Of Minnesota Medical Center, Minneapolis, Minnesota
  - Alamance Regional Medical Center - Cancer Center, Burlington, North Carolina
  - Duke University Medical Center - Morris Cancer Center Clinics, Durham, North Carolina
  - Duke University Medical Center- Department of Medicine Oncology, Durham, North Carolina
  - Duke University Medical Center-Duke Cancer Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke University School Of Medicine, Durham, North Carolina
  - Texas Oncology - PA Collins Building 5th Floor, Dallas, Texas
  - Baylor College Of Medicine (Bcm), Houston, Texas
  - Baylor College of Medicine Breast Center, Houston, Texas
  - Fletcher Allen Healthcare, Burlington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - Fletcher Allen Hospital MCHV Campus, Burlington, Vermont
  - Pharmacist, Investigational Drug Service, Burlington, Vermont
  - Fletcher Allan Health Care, Burlington, Vermont
- Argentina (9):
  - Policlinica Privada Site La Plata S.A., La Plata, Buenos Aires
  - Breast Clinica de la Mama, La Plata, Buenos Aires
  - Policlinica Privada Site, La Plata, Buenos Aires
  - Policlinica Privada Site La Plata S. A., La Plata, Buenos Aires
  - Hospital Italiano Cordoba, Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas, Rosario, Santa Fe Province
  - Centro Oncologico Rosario, Rosario, Santa Fe Province
  - Centro Oncologico De Rosario, Rosario, Santa Fe Province
  - Centro Oncologico, Rosario, Santa Fe Province
- Belgium (3):
  - UZ Gasthuisberg, Medische Oncologie, Leuven
  - UZ Gasthuisberg, Leuven
  - Oncologisch Centrum GZA, Wilrijk
- Brazil (8):
  - Jewish General Hospital, Montreal, QC
  - Instituto Nacional DO Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Cancer - HCII, Santo Cristo, Rio de Janeiro
  - Clínica de Oncologia de porto Alegre Sociedade Simples ltda., Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Das Clinicas Da Faculdade De Medicina Da Universidade De Sao Paulo Instituto Central, São Paulo, São Paulo
  - Centro de Pesquisa em Oncologia - CPO, Porto Alegre
  - Instituto Nacional do Cancer, Rio de Janeiro
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
- Italy (3):
  - Dipartimento di Medicina, Divisione di Oncologia Medica, Istituto Europeo di Oncologia, Milan
  - Divisione di Oncologia, Napoli
  - Uo Oncologia Medica 2 Regione Del Veneto Istituto Oncologico Veneto IRCCS Ospedale Busonera, Padua
- VU University Medical Center, Amsterdam, Netherlands
- Malmö University Hospital, Malmo, Sweden
- United Kingdom (2):
  - St Mary's Hospital NHS Trust, London
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021004&StudyName=Study%20Of%20CP-751%2C871%20In%20Combination%20With%20Exemestane%20In%20Postmenopausal%20Women%20With%20Hormone%20Receptor%20Positive%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871 Plus (+) Exemestane: Participants received CP-751,871 20 milligrams per kilogram (mg/kg) on Day 1 of each 3-week cycle as an intravenous (IV) infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression.
- CP-751,871 + Exemestane/CP-751,871 + Fulvestrant: Participants received CP-751,871 20 mg/kg on Day 1 of each 3-week cycle as an IV infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 4-week cycle in combination with fulvestrant, administered according to the local label and standard clinical practice. Participants continued salvage treatment if safety and clinical benefit were observed for up to a total of 26 cycles or beyond, if there was continued clinical benefit, safety, and tolerability.
- Exemestane: Participants received exemestane 25 mg tablets, by mouth, once daily, until disease progression.
- Exemestane/CP-751,871 + Exemestane: Participants received exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 3-week cycle in combination with exemestane 25 mg tablets, by mouth, once daily, for up to a total of 20 months or beyond if safety and clinical benefit were observed.
Period: Overall Study
Arm/Group | CP-751,871 Plus (+) Exemestane | CP-751,871 + Exemestane/CP-751,871 + Fulvestrant | Exemestane | Exemestane/CP-751,871 + Exemestane
Started | 79 | 36 | 61 | 43
Completed | 42 | 22 | 33 | 23
Not Completed | 37 | 14 | 28 | 20
Not completed — Death | 11 | 4 | 8 | 7
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 6 | 9 | 5
Not completed — Study Terminated by Sponsor | 4 | 0 | 4 | 0
Not completed — Other | 10 | 2 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who started treatment, grouped according to main trial therapy treatment actually received.
Groups:
- CP-751,871 + Exemestane: Participants received CP-751,871 20 mg/kg on Day 1 of each 3-week cycle as an IV infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression could have received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 4-week cycle in combination with fulvestrant, administered according to the local label and standard clinical practice. Participants continued salvage treatment if safety and clinical benefit were observed for up to a total of 26 cycles or beyond, if there was continued clinical benefit, safety, and tolerability.
- Exemestane: Participants received exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression could have received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 3-week cycle in combination with exemestane 25 mg tablets, by mouth, once daily, for up to a total of 20 months or beyond if safety and clinical benefit were observed.
- Total: Total of all reporting groups
Arm/Group | CP-751,871 + Exemestane | Exemestane | Total
Number analyzed (Participants) | 115 | 104 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (10.77) | 62.7 (10.86) | 61.9 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 104 | 219
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was calculated from the time of randomization to either progression of disease, death, or treatment discontinuation because of unsatisfactory therapy results (such as global deterioration of health status). Disease progression was defined as 1 or more of the following: radiographic progression (20 percent [%] increase in measurable lesions, appearance of new lesions or unequivocal progression of evaluable lesions as defined by Response Evaluation Criteria in Solid Tumors [RECIST]); occurrence of new pleural/pericardial effusions or ascites confirmed by positive cytology; persistent hypercalcemia requiring more than 2 IV treatments with bisphosphonates; intervention for any cancer-related events (radiations, surgery) or new symptoms related to tumor growth requiring participant discontinuation; development of brain metastasis; or death for any cause. Median PFS was estimated from the Kaplan-Meier curve. 95% confidence interval (CI) is based on the Brookmeyer and Crowley method.
Time Frame: Baseline, Day 1 of Cycles 2 and 4 and then Day 1 of every 3rd cycle starting at Cycle 7 up to 60 months
Population: Full Analysis Set (FAS): all enrolled participants; grouped by randomized arm, where the first 10 participants enrolled but not randomly assigned to treatment were not included.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CP-751,871 + Exemestane: Participants were assigned to receive CP-751,871 20 mg/kg on Day 1 of each 3-week cycle as an IV infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression.
- Exemestane: Participants were assigned to receive exemestane 25 mg tablets, by mouth, once daily, until disease progression.
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 106 | 103
months | 11.0 [8.1 to 12.9] | 9.2 [7.0 to 13.0]
Statistical Analysis 1: Comparison: CP-751,871 + Exemestane vs Exemestane; Test type: Superiority or Other; p = 0.560, Log Rank; 2-sided p-value from an unstratified log-rank text; Hazard Ratio (HR) = 0.912, 80% CI 2-sided [0.744 to 1.118] — Hazard ratio was based on Cox proportional hazards model

2. Primary Outcome: PFS in Participants With Hemoglobin A1c (HbA1c) Less Than (<) 5.7% at Baseline
Description: PFS was calculated from the time of randomization to either progression of disease, death, or treatment discontinuation because of unsatisfactory therapy results (such as global deterioration of health status). Disease progression was defined as 1 or more of the following: radiographic progression (20% increase in measurable lesions, appearance of new lesions or unequivocal progression of evaluable lesions as defined by RECIST); occurrence of new pleural/pericardial effusions or ascites confirmed by positive cytology; persistent hypercalcemia requiring more than 2 IV treatments with bisphosphonates; intervention for any cancer-related events (radiations, surgery) or new symptoms related to tumor growth requiring participant discontinuation; development of brain metastasis; or death for any cause. Median PFS was estimated from the Kaplan-Meier curve. 95% CI is based on the Brookmeyer and Crowley method.
Time Frame: Baseline, Day 1 of Cycles 2 and 4 and then Day 1 of every 3rd cycle starting at Cycle 7 up to 60 months
Population: FAS; only participants with baseline HbA1c <5.7% were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 39 | 40
months | 13.2 [8.1 to 19.5] | 9.9 [7.0 to 13.6]
Statistical Analysis 1: Comparison: CP-751,871 + Exemestane vs Exemestane; Test type: Superiority or Other; p = 0.331, Log Rank — 2-sided p-value from unstratified log-rank test; Hazard Ratio (HR) = 0.764, 70% CI 2-sided [0.572 to 1.020] — Hazard ratio was based on the Cox proportional hazards model

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD) Maintained for at Least 6 Months
Description: Objective responses were defined using RECIST as CR: disappearance of all target and nontarget lesions. PR: at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the baseline sum LD. Nontarget lesions may persist provided there is no unequivocal progression in these lesions. SD: measurements demonstrating neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as progressive disease (PD) during the first 6 weeks after the start of treatment taking as reference the smallest sum LD since the treatment started. During this time, nontarget lesions may persist provided there is no unequivocal progression in these lesions.
Time Frame: Baseline, Day 1 of Cycles 2 and 4 and then Day 1 of every 3rd cycle starting at Cycle 7 up to 60 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 106 | 103
percentage of participants | 68.9 [59.1 to 77.5] | 64.1 [54.0 to 73.3]
Statistical Analysis 1: Comparison: CP-751,871 + Exemestane vs Exemestane; Test type: Superiority or Other; p = 0.463, Pearson chi-square test; Mean Difference (Net) = 4.790, 95% CI 2-sided [-8.0 to 17.6]

4. Secondary Outcome: Maximum Plasma Concentration of CP-751,871
Time Frame: Predose on Day 1 at Cycles 1, 2, 4, and 5 and 150 days post last dose of CP-751,871 and for salvage therapy, at Day 1 and 150 days post last dose of CP-751,871
Population: The study was terminated early due to strategic reasons and pharmacokinetic (PK) sampling was discontinued by Protocol Amendment 6. Therefore, the analysis was not performed and an incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading.
Groups:
- CP-751,871 + Exemestane: Participants received CP-751,871 20 mg/kg on Day 1 of each 3-week cycle as an IV infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression.
Arm/Group | CP-751,871 + Exemestane
Number analyzed (Participants) | 0

5. Secondary Outcome: Minimum Plasma Concentration of CP-751,871
Time Frame: as for outcome 4
Population: The study was terminated early due to strategic reasons and PK sampling was discontinued by Protocol Amendment 6. Therefore, the analysis was not performed and an incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading.
Arm/Group | CP-751,871 + Exemestane
Number analyzed (Participants) | 0

6. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to the Last Time Point With Quantifiable Concentration
Time Frame: as for outcome 4
Population: as for outcome 5
Arm/Group | CP-751,871 + Exemestane
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Negative Human Anti-Human Antibodies (HAHAs)
Description: Negative human anti-human antibodies were defined as <6.64
Time Frame: Predose on Day 1 of Cycle 1 and at 150 days post last CP-751,871 infusion
Population: All randomized participants who started treatment and who had at least 1 sample submitted for the biomarker; collection of samples for this analysis was stopped after Amendment 6. All samples were negative to HAHA.
Measure: Number; unit: participants
Units Other Than Participants: samples
Arm/Group | CP-751,871 + Exemestane
Number analyzed (Participants) | 37
Number analyzed (samples) | 66
participants | 37

8. Secondary Outcome: Percentage of Participants With Circulating Tumor Cells Expressing Insulin-Like Growth Factor 1 Receptor (IGF-IR)
Time Frame: Predose on Day 1 of Cycle 1
Population: The study was terminated early due to strategic reasons and biomarker sampling was discontinued by Protocol Amendment 6. Therefore, the analysis was not performed and an incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading.
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Serum Markers Relevant to the IGF-1R Pathway
Time Frame: Predose on Day 1 of Cycles 1 and 4 and at end of treatment prior to beginning salvage therapy
Population: as for outcome 8
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 30 (QLQ-C30) Scores
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score equals (=) better level of functioning or greater degree of symptoms.
Time Frame: Predose on Day 1 of each cycle, at the end of treatment and at follow-up, up to 60 months
Population: The study was terminated early secondary to strategic reasons and the questionnaires were discontinued by Protocol Amendment 6. Therefore, the analysis was not performed and an incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading.
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: EORTC QLQ Breast Cancer Module (BR23) Scores
Description: EORTC-QLQ-BR23: included functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions used 4-point Likert scale (1 â€˜Not at Allâ€™ to 4 â€˜Very Muchâ€™). Scores averaged and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Predose on Day 1, at end of treatment, and at Follow-up, up to 60 months
Population: as for outcome 10
Arm/Group | CP-751,871 + Exemestane | Exemestane
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) recorded from informed consent through and including 150 calendar days after the last administration of investigational product. Active reporting period for exemestane/fulvestrant clarified to 28 days after last dose in Amendment 6.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- CP-751,871 + Fulvestrant (After CP-751,871+Exemestane): Participants received CP-751,871 20 mg/kg on Day 1 of each 3-week cycle as an IV infusion in combination with exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 4-week cycle in combination with fulvestrant, administered according to the local label and standard clinical practice. Participants continued salvage treatment if safety and clinical benefit were observed for up to a total of 26 cycles or beyond, if there was continued clinical benefit, safety, and tolerability. Adverse events are presented from the period of time when the participant was receiving salvage therapy treatment only.
- CP-751,871 + Exemestane (After Exemestane): Participants received exemestane 25 mg tablets, by mouth, once daily, until disease progression. Participants who experienced disease progression received salvage therapy with CP-751,871 20 mg/kg on Day 1 of each 3-week cycle in combination with exemestane 25 mg tablets, by mouth, once daily, for up to a total of 20 months or beyond if safety and clinical benefit were observed. Adverse events are presented from the period of time when the participant was receiving salvage therapy treatment only.
Arm/Group | CP-751,871 + Exemestane | CP-751,871 + Fulvestrant (After CP-751,871+Exemestane) | Exemestane | CP-751,871 + Exemestane (After Exemestane)
Serious Adverse Events (participants affected / at risk) | 38/115 | 11/36 | 23/104 | 15/43
Other Adverse Events (participants affected / at risk) | 113/115 | 34/36 | 96/104 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 + Exemestane (N=115) | CP-751,871 + Fulvestrant (After CP-751,871+Exemestane) (N=36) | Exemestane (N=104) | CP-751,871 + Exemestane (After Exemestane) (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Disease progression (General disorders) | 5 | 2 | 4 | 6
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 0 | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Open reduction of fracture (Surgical and medical procedures) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 + Exemestane (N=115) | CP-751,871 + Fulvestrant (After CP-751,871+Exemestane) (N=36) | Exemestane (N=104) | CP-751,871 + Exemestane (After Exemestane) (N=43)
Anaemia (Blood and lymphatic system disorders) | 8 | 3 | 9 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 10 | 41 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 6 | 18 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 11 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 3
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 41 | 12 | 4 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 10 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 5 | 15 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 2 | 9 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 7 | 16 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2
Hot flush (Vascular disorders) | 13 | 5 | 25 | 7
Hypertension (Vascular disorders) | 14 | 3 | 4 | 3
Deafness (Ear and labyrinth disorders) | 7 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 2 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 6 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 7 | 0 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 8 | 3 | 2 | 0
Dry eye (Eye disorders) | 7 | 1 | 4 | 1
Eye pain (Eye disorders) | 3 | 2 | 0 | 1
Lacrimation increased (Eye disorders) | 6 | 1 | 3 | 1
Vision blurred (Eye disorders) | 7 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 3 | 11 | 3
Abdominal pain upper (Gastrointestinal disorders) | 9 | 1 | 6 | 3
Constipation (Gastrointestinal disorders) | 29 | 8 | 16 | 7
Diarrhoea (Gastrointestinal disorders) | 37 | 8 | 22 | 12
Dry mouth (Gastrointestinal disorders) | 15 | 2 | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 9 | 4 | 9 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 2 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 6 | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 35 | 8 | 19 | 15
Stomatitis (Gastrointestinal disorders) | 8 | 4 | 0 | 1
Toothache (Gastrointestinal disorders) | 10 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 23 | 4 | 6 | 7
Asthenia (General disorders) | 17 | 3 | 13 | 8
Chest pain (General disorders) | 8 | 2 | 8 | 1
Fatigue (General disorders) | 35 | 11 | 33 | 16
Influenza like illness (General disorders) | 6 | 1 | 2 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 10 | 3
Pain (General disorders) | 7 | 2 | 8 | 6
Pyrexia (General disorders) | 11 | 1 | 5 | 1
Palpitations (Cardiac disorders) | 7 | 1 | 6 | 0
Cystitis (Infections and infestations) | 6 | 0 | 5 | 3
Nasopharyngitis (Infections and infestations) | 13 | 0 | 9 | 0
Sinusitis (Infections and infestations) | 6 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 0 | 7 | 2
Urinary tract infection (Infections and infestations) | 21 | 3 | 8 | 8
Alanine aminotransferase increased (Investigations) | 9 | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 6 | 2 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 15 | 3 | 2 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 3
Weight decreased (Investigations) | 34 | 10 | 5 | 14
Dysuria (Renal and urinary disorders) | 11 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 41 | 13 | 13 | 13
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 50 | 9 | 4 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 3
Amnesia (Nervous system disorders) | 3 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 21 | 3 | 13 | 6
Dysgeusia (Nervous system disorders) | 21 | 2 | 1 | 7
Headache (Nervous system disorders) | 29 | 7 | 23 | 13
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 6 | 3 | 5 | 1
Anxiety (Psychiatric disorders) | 8 | 2 | 4 | 3
Confusional state (Psychiatric disorders) | 7 | 2 | 3 | 2
Depression (Psychiatric disorders) | 13 | 4 | 15 | 12
Insomnia (Psychiatric disorders) | 13 | 2 | 15 | 5
Breast pain (Reproductive system and breast disorders) | 6 | 2 | 10 | 5
Pelvic pain (Reproductive system and breast disorders) | 4 | 2 | 3 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 6 | 3 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 4 | 17 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 6 | 14 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 3 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 2 | 8 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 2 | 3 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 25 | 11 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 2 | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 7 | 0 | 4 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No